CLINICAL TRIAL: NCT07249125
Title: A Prospective Registry Study Evaluating the Safety and Quality of Life of Three Treatment Strategies - Surgical Resection, Thermal Ablation, and Active Surveillance - for Patients With Low-Risk Papillary Thyroid Microcarcinoma
Brief Title: Safety and Quality of Life of Three Treatment Strategies for Low-Risk Papillary Thyroid Microcarcinoma
Acronym: PTMC-3S
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20252532-C-1
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Papillary Thyroid Microcarcinoma
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical Resection: Participants undergo standard thyroid surgery (lobectomy or total thyroidectomy) for low-risk papillary thyroid microcarcinoma. Outcomes on safety, complications, and postoperative quality of life are collected prospectively.
- Thermal Ablation: Participants receive minimally invasive thermal ablation, such as radiofrequency or microwave ablation, for papillary thyroid microcarcinoma. Data include procedural safety, ablation completeness, and patient-reported quality of life.
- Active Surveillance: Participants choose active surveillance instead of immediate intervention. Regular follow-up with ultrasound and clinical assessment is conducted to monitor tumor progression, safety events, and quality of life over time.

SUMMARY:
This is a prospective observational patient registry study designed to evaluate the safety and quality of life associated with three treatment strategies for patients diagnosed with low-risk papillary thyroid microcarcinoma (PTMC): surgical resection, thermal ablation, and active surveillance.

The study aims to collect standardized, real-world clinical data from participating centers. Patients will receive one of the three treatment strategies according to clinical judgment and personal preference. The study team will prospectively follow participants to record safety events, disease progression, and patient-reported quality of life outcomes.

By comparing the outcomes among the three treatment groups, this registry seeks to provide evidence to support personalized and evidence-based decision-making for the management of low-risk PTMC.

ELIGIBILITY:
Inclusion Criteria:

* A single papillary thyroid carcinoma (PTC) lesion with a maximum diameter ≤ 1 cm confirmed by imaging.
* No evidence of extrathyroidal extension on imaging studies.
* No clinical or radiologic evidence of cervical lymph node metastasis.
* No evidence of distant metastasis.
* Histopathological confirmation of papillary thyroid carcinoma.
* The patient has provided written informed consent and agrees to select one of the predefined management strategies (surgical resection, thermal ablation, or active surveillance).

Exclusion Criteria:

* Ultrasound-confirmed tumor with a maximum diameter > 1 cm.
* Imaging findings (ultrasound/CT/MRI) suggestive of extrathyroidal extension.
* Tumor located adjacent to critical structures (e.g., trachea, esophagus, or recurrent laryngeal nerve) with possible invasion risk.
* History of thyroidectomy, radiofrequency/microwave/laser ablation, or radioactive iodine therapy.
* Failure to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with low-risk papillary thyroid microcarcinoma (maximum diameter ≤1 cm), with no evidence of extrathyroidal extension, lymph node metastasis, or distant metastasis, who choose one of three management strategies: surgical resection, thermal ablation, or active surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 1630 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2038-12-31 (Estimated); Study Completion 2039-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of lymph node metastasis confirmed by imaging and fine-needle aspiration within 10 years | 10 years
  The proportion of participants who show radiologic evidence of lymph node metastasis confirmed by fine-needle aspiration during 10 years of follow-up.

SECONDARY OUTCOMES:
Rate of lymph node metastasis confirmed by imaging and fine-needle aspiration within 5 years | 5 years
  The proportion of participants with imaging findings suggestive of lymph node metastasis confirmed by fine-needle aspiration at 5 years.
Proportion of nodules with ≥3 mm increase in maximal diameter on ultrasound within 5 years (Active Surveillance group) | 5 years
  Among participants in the active surveillance group, the proportion of thyroid nodules showing an ultrasound-measured increase of at least 3 mm in maximal diameter within 5 years of follow-up.
Proportion of nodules with ≥3 mm increase in maximal diameter on ultrasound within 10 years (Active Surveillance group) | 10 years
  Among active surveillance participants, the proportion of thyroid nodules showing an ultrasound-measured increase of 3 mm or more in maximal diameter within 10 years.
Overall survival rate at 10 years | 10 years
  The proportion of participants who remain alive at 10 years from baseline, regardless of disease status or treatment modality.
Conversion rate from active surveillance to surgery | Up to 10 years
  The proportion of participants initially managed with active surveillance who undergo surgical intervention during the study period.
Quality of life scores at 1, 3, 5, and 10 years | 1, 3, 5, and 10 years
  Changes in patient-reported quality of life over time, evaluated using the Fear of Progression Questionnaire-Short Form (FoP-Q-SF) and the Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QoL).

OTHER OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Throughout the 10-year follow-up period
  Number and percentage of participants experiencing any study-related adverse events or serious adverse events, collected throughout the study and categorized by severity and relationship to treatment type.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request after publication of the main results. Data will be shared with qualified researchers with a methodologically sound proposal, subject to approval by the study steering committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after main publication; available for at least 5 years thereafter.
Access Criteria: Researchers may request access through the corresponding author by submitting a proposal and a data use agreement.